CLINICAL TRIAL: NCT02495168
Title: A Randomized, Blinded, Parallel Group, Placebo-Controlled, Multiple Dose, Multicenter, Multinational Study to Compare the Therapeutic Equivalence of a Budesonide 80 μg/Formoterol Fumarate Dihydrate 4.5 μg Inhalation Aerosol (Manufactured by Catalent for Watson Laboratories Inc.) to Symbicort® (Budesonide 80 μg/Formoterol Fumarate Dihydrate 4.5 μg Inhalation Aerosol) (Manufactured by AstraZeneca) in Adolescent and Adult Patients With Asthma
Brief Title: Randomized, Placebo-Controlled, Multidose, Study Comparing Generic Budesonide/Formoterol Fumarate Dihydrate to Symbicort® in Asthmatic Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT-2015-075-0AA
Record Dates: First submitted 2015-07-01; First posted 2015-07-13 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Generic Budesonide/Formoterol Fumarate Dihydrate (Experimental): After a 2-week Run-in Period of administering 2 inhalations twice daily via a generic placebo pMDI device, participants will administer 2 inhalations twice daily via a generic budesonide/formoterol fumarate dihydrate (80 μg/4.5 μg) pMDI for up to 50 days.
  Interventions: Drug: Generic Budesonide/Formoterol Fumarate Dihydrate
- Symbicort (Budesonide/Formoterol Fumarate Dihydrate) (Active Comparator): After a 2-week Run-in Period of administering 2 inhalations twice daily via a generic placebo pMDI device, participants will administer 2 inhalations twice daily via a Symbicort budesonide/formoterol fumarate dihydrate (80 μg/4.5 μg) pMDI for up to 50 days.
  Interventions: Drug: Symbicort® (Budesonide/Formoterol Fumarate Dihydrate)
- Placebo (Placebo Comparator): After a 2-week Run-in Period of administering 2 inhalations twice daily via a generic placebo pMDI device, participants will administer 2 inhalations twice daily via a generic placebo pMDI for up to 50 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Generic Budesonide/Formoterol Fumarate Dihydrate — Oral inhalation, generic formulation of the brand-name product.
  Arms: Generic Budesonide/Formoterol Fumarate Dihydrate
Drug: Symbicort® (Budesonide/Formoterol Fumarate Dihydrate) — Oral inhalation, brand-name product.
  Other Names: Symbicort Turbohaler®
  Arms: Symbicort (Budesonide/Formoterol Fumarate Dihydrate)
Drug: Placebo — Oral inhalation, no active ingredient.
  Arms: Placebo

SUMMARY:
This study has a randomized multiple-dose, placebo-controlled, parallel group design consisting of a 2-week open placebo Run-in Period followed by a 6-week Treatment Period with placebo, test product (budesonide 80 microgram [μg]/formoterol fumarate dihydrate 4.5 μg), or reference product (Symbicort® inhalation aerosol).

DETAILED DESCRIPTION:
This is a pivotal trial that will examine the therapeutic equivalence of a new generic fixed-dose combination product containing budesonide 80 μg/formoterol fumarate dihydrate 4.5 μg and reference listed drug (RLD) Symbicort® inhalation aerosol in adult participants with chronic but stable asthma as defined in National Asthma Education and Prevention Program Expert Panel Report 3 (NAEPP 3) guidelines. To ensure adequate study sensitivity, the test and reference products should both be statistically superior to placebo (p<0.05) with regard to the bioequivalent study primary endpoints. Participants will be provided a generic placebo pressurized metered-dose inhaler (pMDI) device for use during the 2-week Run-in Period for device training.

ELIGIBILITY:
Inclusion criteria:

1. Adolescent and adult male or female participants (≥12 and ≤75 years of age).
2. Female participants must not be lactating or pregnant at Screening, as documented by a negative serum pregnancy test with a minimum sensitivity of 25 international unit/liter (IU/L) or equivalent units of beta-human chorionic gonadotropin (β-hCG) at Screening.
3. Women of childbearing potential (WOCBP) and female partners (WOCBP) of male participants participating in the study, must commit to consistent and correct use of an acceptable method of birth control (at the Investigator's discretion) throughout the study and for 30 days after study drug discontinuation.
4. Male participants and male partners of female participants (WOCBP) must commit to consistent and correct use of an acceptable method of birth control (at the Investigator's discretion) throughout the study and for 30 days after the study drug discontinuation.
5. Diagnosed with asthma as defined by the NAEPP 3 at least 6 months prior to Screening. If the participant is new to the study site, the Investigator must confirm the participant's asthma diagnosis. Acceptable means include either medical records or pharmacy records.
6. Moderate to severe asthma with a pre-bronchodilator forced expiratory volume in 1 second (FEV1) of ≥45% and ≤85% of the predicted normal value during measured at least 6 hours after short-acting β agonist (SABA) and at least 24 hours after the last dose of long-acting β agonist (LABA) at Screening and prior to randomization on Day 1.
7. Currently non-smoking, negative for urine cotinine at Screening, having not used tobacco products (that is, cigarettes, cigars, pipe tobacco, and electronic cigarettes) within the past year, and had ≤10 pack-years of historical use.
8. Body mass index (BMI) between 18 to 40 (inclusive) for participants ≥18 years old. For adolescent participants 12 to 17 years old, BMI between 15 to 40 inclusive (in accordance with the BMI range typical for the age).
9. ≥15% and ≥0.20 L reversibility of FEV1 within 30 minutes following 360 μg (4 puffs) of albuterol (400 μg salbutamol) inhalation (pMDI). If the participant achieves <15%, but ≥10% reversibility at the Screening, the site may instruct the participant to hold LABA and/or inhaled corticosteroids (ICS) and return up to 7 days later for a repeat test. Only 1 repeat of the Screening spirometry test (to retest reversibility) is allowed.
10. Able to perform valid and reproducible spirometry results per American Thoracic Society/European Respiratory Society (ATS/ERS) standards at Screening.
11. Able to inhale study drug properly.
12. Willing to discontinue asthma medications (ICS and LABAs) during the Run-in Period and for the remainder of the study.
13. Able to replace current regularly scheduled SABAs with albuterol/salbutamol inhaler for use only on as needed basis for the duration of the study (participants should be able to withhold all inhaled SABAs for at least 6 hours prior to lung function assessments on study visits).
14. Able to continue the following medications without a significant adjustment of dosage, formulation, dosing interval for the duration of the study, and judged able by the Investigator to withhold them for the specified minimum time intervals prior to each clinic visit, if applicable:

    1. Short-acting forms of theophylline: 12 hours.
    2. Twice-a-day controlled-release forms of theophylline: 24 hours.
    3. Once-a-day controlled-release forms of theophylline: 36 hours.
15. Able to discontinue the following medications for the specified minimum time intervals prior to the Run-in Period and for the remainder of the study, if applicable:

    1. Oral corticosteroids for 30 days.
    2. Parenteral corticosteroids for 30 days.
    3. Oral (not inhaled) SABAs for 24 hours.
16. Clinical laboratory tests (clinical chemistry, hematology, and urinalysis) and 12-lead electrocardiogram (ECG) conducted at Screening within normal limits or abnormal but not clinically significant to the Investigator. The QTc should be calculated using Bazett's formula.
17. Willing to give written informed consent/assent, and willing and able to follow the study rules and procedures.
18. Stable on chronic asthma treatment regimen for at least 4 weeks prior to enrollment.
19. Ability to perform forced expiratory assessments according to ATS standards.

Randomization eligibility criteria:

1. Baseline pre-bronchodilator FEV1 should be ≥45% and ≤85% of predicted normal value and not vary by more than ±20% from Screening FEV1 value.
2. Compliance during the Run-in Period of at least 75% based on electronic Diary entries is required for a participant to qualify for randomization. Compliance with the run-in placebo treatment must be between 75% and 125%.
3. Documented total asthma symptom score of ≥1 for at least 2 days during the Run-in Period.

Exclusion criteria:

1. Life-threatening asthma, defined as a history of asthma episode(s) requiring intubation, and/or associated with hypercapnea, respiratory arrest or hypoxic seizures, asthma-related syncopal episode(s), or hospitalizations within the past year or during the Run-in Period.
2. Exercise-induced asthma as the only asthma-related diagnosis.
3. Evidence or history of clinically significant disease or abnormality including congestive heart failure, uncontrolled hypertension, uncontrolled coronary artery disease, myocardial infarction, or cardiac dysrhythmia. In addition, historical or current evidence of significant hematologic, hepatic, neurologic, psychiatric, renal, or other diseases that in the opinion of the Investigator would put the participant at risk through study participation or would affect the study analyses if the disease exacerbated during the study. Participants with well-controlled hypertension, diabetes or hypercholesterolemia are not excluded as long as their medication does not interfere with the study.
4. Any other clinically significant pulmonary disease except for asthma, including chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, bronchiectasis, chronic bronchitis, emphysema, active pulmonary tuberculosis, pulmonary carcinoma, pulmonary fibrosis, or pulmonary hypertension. In addition, obstructive sleep apnea warranting a prescription for continuous or biphasic positive airway pressure (continuous positive airway pressure [CPAP] or bilevel positive airway pressure [BiPAP]).
5. Participants who required systemic corticosteroids (for any reason) within the past 4 weeks.
6. Participants with hypersensitivity to any sympathomimetic drug (for example, formoterol, albuterol/salbutamol, or salmeterol) or any inhaled, intranasal, or systemic corticosteroid therapy.
7. Participants taking medication(s) (either daily or as needed) with the potential to affect the course of asthma or to interact with sympathomimetic amines, for example:

   1. Oral β-blockers.
   2. Strong cytochrome P450 3A4 inhibitors (for example, ritonavir).
   3. Monoclonal antibodies/Biologic agents which may affect the course of asthma (such as mepolizumab, reslizumab, lebrikizumab, and others).
8. Viral or bacterial, upper or lower respiratory tract infection or sinus or middle ear infection within 2 weeks prior to Screening or during the Run-in Period.
9. Factors (for example, infirmity, disability or geographic location) that the Investigator feels would likely limit the participant's compliance with the study protocol or scheduled clinic visits.
10. Anti-Immunoglobulin E (IgE) (such as omalizumab) use within the 6 months prior to screening.
11. History of alcohol or drug abuse within the last 6 months.
12. A positive urine drug screen at Screening. Exceptions are made for a positive urine drug screen at Screening for opiates or stimulants if there is a documented prescription with supporting medical history and diagnosis, and the Principal Investigator assesses there are no safety concerns with participant participation. Screened participants with a urine drug screen positive for marijuana/tetrahydrocannabinol are not eligible for study participation, without exceptions. Repeat drug screening is not allowed.
13. Have received any other investigational treatment within 30 days (or within 5 terminal half-lives of the investigational drug whichever is longer) of Screening or plans to receive investigational treatment within 30 days after the study is completed.
14. Be an Investigator, employee, or otherwise be directly affiliated with the study site, Watson Laboratories Inc. and affiliates, or service provider involved in the study including being an immediate family member of an Investigator or site employee (that is, spouse, parent, child, or sibling), whether biological or legally adopted or in foster care.
15. Non-compliance with the study requirements, rules, and procedures.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1714 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Site 100, Surprise, Arizona
  - Site 101, Huntington Beach, California
  - 111, San Jose, California
  - 114, Centennial, Colorado
  - 104, Hialeah, Florida
  - 103, Miami, Florida
  - 105, Miami, Florida
  - 107, Miami, Florida
  - 106, Bozeman, Montana
  - 113, Bellevue, Nebraska
  - 112, Cincinnati, Ohio
  - 108, Edmond, Oklahoma
  - 115, Eugene, Oregon
  - 116, Medford, Oregon
  - 110, Rock Hill, South Carolina
  - 109, Smyrna, Tennessee
  - 102, Waco, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (N=1714) were provided a generic placebo pressurized metered dose inhaler (pMDI) device for use during a 2-week Run-in Period for device training. Then, qualified participants (N=1147) were randomly assigned to treatment on a 4:4:1 ratio of generic budesonide/formoterol fumarate dihydrate, Symbicort, or Placebo, respectively.
Groups:
- Generic Budesonide/Formoterol Fumarate Dihydrate: After a 2-week Run-in Period of administering 2 inhalations twice daily via a generic placebo pMDI device, participants administered 2 inhalations twice daily via a generic budesonide/formoterol fumarate dihydrate (80 microgram [μg]/4.5 μg) pMDI for up to 50 days.
- Symbicort (Budesonide/Formoterol Fumarate Dihydrate): After a 2-week Run-in Period of administering 2 inhalations twice daily via a generic placebo pMDI device, participants administered 2 inhalations twice daily via a Symbicort budesonide/formoterol fumarate dihydrate (80 μg/4.5 μg) pMDI for up to 50 days.
- Placebo: After a 2-week Run-in Period of administering 2 inhalations twice daily via a generic placebo pMDI device, participants administered 2 inhalations twice daily via a generic placebo pMDI for up to 50 days.
Period: Overall Study
Arm/Group | Generic Budesonide/Formoterol Fumarate Dihydrate | Symbicort (Budesonide/Formoterol Fumarate Dihydrate) | Placebo
Started | 504 | 516 | 127
Safety Population (Randomized participants who received at least 1 dose of study drug during Treatment Period) | 501 | 514 | 126
Modified Intent-to-Treat Population (Participants in Safety Population with no major inclusion/exclusion deviations, enrolled only once) | 468 | 478 | 111
Day1 Per-protocol Set (D1PPS) Population (mITT Population, no major protocol violations that impacted analysis of the Day 1 primary endpoint) | 437 | 437 | 99
Day 42 (D42PPS) Population (mITT Population, no major protocol violations that impacted analysis of the Day 42 primary endpoint) | 382 | 383 | 88
Completed | 466 | 462 | 110
Not Completed | 38 | 54 | 17
Not completed — Other than Specified | 18 | 22 | 5
Not completed — Did not Complete Final Visit On Time | 4 | 3 | 2
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Lost to Follow-up | 10 | 6 | 1
Not completed — Withdrawal by Subject | 1 | 4 | 2
Not completed — Protocol Violation | 0 | 10 | 1
Not completed — Adverse Event | 4 | 8 | 3
Not completed — Lack of Efficacy | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Randomized participants who received at least 1 dose of study drug during Treatment Period (Safety Population).
Groups:
- Generic Budesonide/Formoterol Fumarate Dihydrate: After a 2-week Run-in Period of administering 2 inhalations twice daily via a generic placebo pMDI device, participants administered 2 inhalations twice daily via a generic budesonide/formoterol fumarate dihydrate (80 μg/4.5 μg) pMDI for up to 50 days.
- Total: Total of all reporting groups
Arm/Group | Generic Budesonide/Formoterol Fumarate Dihydrate | Symbicort (Budesonide/Formoterol Fumarate Dihydrate) | Placebo | Total
Number analyzed (Participants) | 501 | 514 | 126 | 1141
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (15.39) | 43.9 (15.56) | 41.5 (15.88) | 43.1 (15.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 299 | 292 | 70 | 661
  Male | 202 | 222 | 56 | 480
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 171 | 180 | 48 | 399
  Not Hispanic or Latino | 330 | 334 | 78 | 742
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 9 | 11 | 5 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 90 | 86 | 23 | 199
  White | 402 | 410 | 97 | 909
  More than one race | 0 | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Forced Expiratory Volume in 1 Second (FEV1) [Mean (Standard Deviation); unit: liters] — FEV1 was measured using spirometry in accordance with the American Thoracic Society/European Respiratory Society (ATS/ERS) consensus guidelines. Data collected at pre-inhalation at Baseline is presented. Population: Participants who received at least 1 dose of study drug, no major inclusion/exclusion violations, and enrolled in the study only once (Modified Intent-to-Treat [mITT] Population) and with evaluable FEV1 data.
  liters
    number analyzed (Participants) | 466 | 476 | 111 | 1053
    (all) | 2.113 (0.5524) | 2.083 (0.5400) | 2.136 (0.5975) | 2.102 (0.5515)

OUTCOME MEASURES:

1. Primary Outcome: Equivalence Analysis of Area Under the Serial FEV1-Time Effect Curve From Time 0 to 12 Hours (FEV1 Area Under Curve [AUC0-12]) on the First Day of Treatment
Description: FEV1 was measured using spirometry in accordance with the ATS/ERS consensus guidelines. Baseline-adjusted area under the serial FEV1-time curve was calculated from Time 0 to 12 hours on the first day of the Treatment Period (Day 1). FEV1 AUC0-12 was calculated from baseline-adjusted values using the linear trapezoidal method. The calculation assumed that at time of dosing (Time 0) the baseline adjusted FEV1 was also 0. The calculation proceeded over all available post-dose FEV1 assessments on Day 1 (including unscheduled time points, if any) using actual elapsed time from dosing. FEV1 baseline defined as the average of predose FEV1 values obtained on Day 1. If some of these values were missing, the average was calculated using the available values, however, a minimum of 2 predose FEV1 values were required; participants who had only 1 or no predose FEV1 measurements on Day 1 would have their FEV1 baseline missing, and the participant was to be excluded from analysis.
Time Frame: 0 to 12 hours on Day 1
Population: Randomized participants who received at least 1 dose of study drug, no major inclusion/exclusion violations, enrolled in the study only once, and no major protocol violations that impacted analysis of the Day 1 FEV1 AUC (D1PPS Population).
Measure: Mean (Standard Deviation); unit: Liter*hour (Lh)
Arm/Group | Generic Budesonide/Formoterol Fumarate Dihydrate | Symbicort (Budesonide/Formoterol Fumarate Dihydrate) | Placebo
Number analyzed (Participants) | 437 | 437 | 99
Liter*hour (Lh) | 3.637 (3.2532) | 3.584 (2.9913) | 1.460 (3.3183)
Statistical Analysis 1: Comparison: Generic Budesonide/Formoterol Fumarate Dihydrate vs Symbicort (Budesonide/Formoterol Fumarate Dihydrate); Test type: Equivalence — To show the clinical equivalence, an analysis of covariance (ANCOVA) model was fit on the participants from the generic budesonide/formoterol fumarate and Symbicort groups only, with the endpoint as outcome and treatment, study site and treatment by site interaction as fixed effects and FEV1 baseline value as covariate. If the treatment-by-site interaction factor was not significant at the 0.05 level, the model was to be rerun without the interaction term; Test/Referece LS Mean Ratio = 101.9, 90% CI 2-sided [92.7 to 111.9] — Fieller's formula was applied to calculate the 90% confidence interval (CI) for the generic budesonide/formoterol fumarate and Symbicort LS mean ratio; covariance between treatment means was assumed to be 0

2. Primary Outcome: Superiority Analysis of Area Under the Serial FEV1-Time Effect Curve From Time 0 to 12 Hours (FEV AUC0-12) on the First Day of Treatment
Description: as for outcome 1
Time Frame: 0 to 12 hours on Day 1
Population: Randomized participants who received at least 1 dose of study drug, no major inclusion/exclusion violations, and enrolled in the study only once (mITT Population) and with evaluable FEV1 AUC data.
Measure: Mean (Standard Deviation); unit: Lh
Arm/Group | Generic Budesonide/Formoterol Fumarate Dihydrate | Symbicort (Budesonide/Formoterol Fumarate Dihydrate) | Placebo
Number analyzed (Participants) | 468 | 478 | 111
Lh | 3.630 (3.2528) | 3.573 (2.9960) | 1.449 (3.3033)
Statistical Analysis 1: Comparison: Generic Budesonide/Formoterol Fumarate Dihydrate vs Placebo; LS means difference and p-value from ANCOVA model with treatment and site as fixed effects, baseline FEV1 as covariate and endpoint as outcome on generic budesonide/formoterol fumarate dihydrate and Placebo participants only; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = 2.334, 95% CI 2-sided [1.673 to 2.996]
Statistical Analysis 2: Comparison: Symbicort (Budesonide/Formoterol Fumarate Dihydrate) vs Placebo; LS means difference and p-value from ANCOVA model with treatment and site as fixed effects, baseline FEV1 as covariate and endpoint as outcome on Symbicort and Placebo participants only; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = 2.606, 95% CI 2-sided [1.939 to 3.273]

3. Primary Outcome: Equivalence Analysis of Baseline-Adjusted Average Predose FEV1 at End of Treatment
Description: FEV1 was measured using spirometry in accordance with the ATS/ERS consensus guidelines. Average predose FEV1 at End of Treatment defined as the average of all predose assessments on Day 42. If a participant had no predose assessment on Day 42, the average of all available predose assessments on the last day (for example, Early Termination visit [up to Day 50]) when at least 1 predose FEV1 assessments was available was imputed, if the participant discontinued due to lack of efficacy, otherwise there was no imputation. Baseline was defined as the average of at least 2 predose FEV1 values obtained on Day 1. The endpoint of baseline-adjusted predose FEV1 at end of treatment was calculated as follows: [FEV1 at end of treatment] - [Baseline FEV1].
Time Frame: Day 1 up to Day 50
Population: Randomized participants who received at least 1 dose of study drug, no major inclusion/exclusion violations, enrolled in the study only once, and no major protocol violations that impacted analysis of the Day 42 FEV1 AUC (D42PPS Population).
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Generic Budesonide/Formoterol Fumarate Dihydrate | Symbicort (Budesonide/Formoterol Fumarate Dihydrate) | Placebo
Number analyzed (Participants) | 382 | 383 | 88
liters | 0.278 (0.3306) | 0.283 (0.3241) | 0.094 (0.3298)
Statistical Analysis 1: Comparison: Generic Budesonide/Formoterol Fumarate Dihydrate vs Symbicort (Budesonide/Formoterol Fumarate Dihydrate); Test type: Equivalence — To show the clinical equivalence, an ANCOVA model was fit on the participants from the generic budesonide/formoterol fumarate and Symbicort groups only, with the endpoint as outcome and treatment, study site and treatment-by site interaction as fixed effects and FEV1 baseline value as covariate. If the treatment-by-site interaction factor was not significant at the 0.05 level, the model was to be rerun without the interaction term; Test/Reference LS Mean Ratio = 99.8, 90% CI 2-sided [87.0 to 114.5] — Fieller's formula was applied to calculate the 90% CI for the generic budesonide/formoterol fumarate and Symbicort LS mean ratio; covariance between treatment means was assumed to be 0

4. Primary Outcome: Superiority Analysis of Baseline-Adjusted Average Predose FEV1 at End of Treatment
Description: as for outcome 3
Time Frame: Day 1 up to Day 50
Population: Randomized participants who received at least 1 dose of study drug, no major inclusion/exclusion violations, and enrolled in the study only once (mITT Population) and with evaluable baseline-adjusted average predose FEV1 data.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Generic Budesonide/Formoterol Fumarate Dihydrate | Symbicort (Budesonide/Formoterol Fumarate Dihydrate) | Placebo
Number analyzed (Participants) | 468 | 478 | 111
liters | 0.269 (0.3238) | 0.277 (0.3156) | 0.124 (0.3673)
Statistical Analysis 1: Comparison: Generic Budesonide/Formoterol Fumarate Dihydrate vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = 0.159, 95% CI 2-sided [0.093 to 0.226]
Statistical Analysis 2: Comparison: Symbicort (Budesonide/Formoterol Fumarate Dihydrate) vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = 0.164, 95% CI 2-sided [0.099 to 0.229]

ADVERSE EVENTS:
Time Frame: First day of the Treatment Period (Day 1) up to Day 72
Description: Randomized participants who received at least 1 dose of study drug during Treatment Period (Safety Population).
Arm/Group | Generic Budesonide/Formoterol Fumarate Dihydrate | Symbicort (Budesonide/Formoterol Fumarate Dihydrate) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/501 | 0/514 | 0/126
Serious Adverse Events (participants affected / at risk) | 3/501 | 2/514 | 1/126
Other Adverse Events (participants affected / at risk) | 70/501 | 79/514 | 15/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Generic Budesonide/Formoterol Fumarate Dihydrate (N=501) | Symbicort (Budesonide/Formoterol Fumarate Dihydrate) (N=514) | Placebo (N=126)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/299 | 0/292 | 0/70 — This is a sex-specific adverse event that only affects female participants.
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Generic Budesonide/Formoterol Fumarate Dihydrate (N=501) | Symbicort (Budesonide/Formoterol Fumarate Dihydrate) (N=514) | Placebo (N=126)
Sinusitis (Infections and infestations) | 0 | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 12 | 8 | 3
Viral upper respiratory tract infection (Infections and infestations) | 10 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 6 | 0
Headache (Nervous system disorders) | 5 | 11 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Adverse drug reaction (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 1 | 0
Hernia pain (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0 | 0
Body tinea (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 2 | 0
Laryngitis (Infections and infestations) | 0 | 1 | 0
Otitis externa (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1/299 | 0/292 | 0/70 — This is a sex-specific adverse event that only affects female participants.
Arthropod sting (Injury, poisoning and procedural complications) | 2 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Neck injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Antinuclear antibody positive (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood glucose decreased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Glucose urine (Investigations) | 0 | 1 | 0
Glucose urine present (Investigations) | 2 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0
Protein urine present (Investigations) | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0
Glycosuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Bunion operation (Surgical and medical procedures) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT02495168/SAP_000.pdf
  • Study Protocol (2017-02-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT02495168/Prot_001.pdf